CLINICAL TRIAL: NCT05001464
Title: Evaluation of Reliability and Validity of Reflectance Pulse Oximeter in Screening Children With Obstructive Sleep Apnea
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, LI-HONG SUN, Researcher, Guangzhou Institute of Respiratory Disease
Other Study IDs: PP of GIRD
Record Dates: First submitted 2021-07-01; First posted 2021-08-12 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Apnea, Obstructive
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Reflectance Pulse Oximeter: The participants wear reflectance pulse oximeter for continuous monitoring when carrying out PSG . Oxygen desaturation index (ODI), average blood oxygen saturation, minimum blood oxygen saturation, percentage of blood oxygen saturation less than 90% in the whole recording time (TS90%), fastest heart rate, slowest heart rate and average heart rate are recorded by reflectance pulse oximeter.
  Interventions: Device: reflectance pulse oximeter

INTERVENTIONS:
Device: reflectance pulse oximeter — Wearing reflectance pulse oximeter at the same time on the night of PSG examination

SUMMARY:
Polysomnography (PSG) has some disadvantages, such as time-consuming, effort-consuming, long appointment time and high cost. During PSG examination, multiple sensors need to be placed in the patient's head, face, neck, chest and limbs, and sensors are needed to monitor data throughout the night. It is difficult for young children to cooperate, and it is easy to fail due to inaccurate sensor signal acquisition. PSG examination may miss diagnosis or underestimate the disease due to the first night effect. Based on the above reasons, the application of PSG in clinic, especially in pediatric patients is limited. The reflective optical path detection can be used to measure the peripheral blood oxygen saturation in the flat part of human skin. The investigators intend to use a reflectance pulse oximeterto evaluate its reliability and validity in the diagnosis of OSA in children at the same time as PSG.

DETAILED DESCRIPTION:
During PSG examination, the participants wear reflectance pulse oximeter for continuous monitoring. Use PSG to record EEG, oculogram, chin electromyography, body movement, chest and abdomen movement, nose and mouth airflow, snoring, electrocardiogram, blood oxygen saturation and finger pulse monitoring. The effective monitoring time should be at least 6 hours. Oxygen desaturation index (ODI), average blood oxygen saturation, minimum blood oxygen saturation, percentage of blood oxygen saturation less than 90% in the whole recording time (TS90%), fastest heart rate, slowest heart rate and average heart rate are recorded by reflectance pulse oximeter. To compare the effective time (TST), the total number of hypoxemia events, the coincidence rate of comparing each hypoxemia event, identifying OSA, and identifying moderate and severe OSA by PSG and reflectance pulse oximeter.

ELIGIBILITY:
Inclusion Criteria:

1. Snoring more than 3 nights per week in the last month
2. Pediatric sleep questionnaires score ≥ 0.33

Exclusion Criteria:

1. Acute exacerbation of asthma
2. Pulmonary infection
3. Heart disease

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 1. With the consent of the guardian, children who are scheduled to undergo PSG examination because of suspected OSA.
  2. There is no serious dysfunction of heart, lung, liver and kidney.
  3. Willing to participate in this project and sign the informed consent form.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Coincidence rate of total number of oxygen reduction events | 1 night
  The ratio of the number of oxygen reduction events recorded by reflectance pulse oximeter consistent with PSG to the total oxygen reduction events of PSG

CONTACTS AND LOCATIONS:
Overall Officials: Jinping Zheng, Professor, Principal Investigator — Guangzhou Institute of Respiratory Health
Locations (1):
- 151 Yanjiang Road, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided